CLINICAL TRIAL: NCT00114296
Title: A Pilot Study to Evaluate the Effects of Omega-3 Fatty Acids on Intermediate Markers of Breast Cancer
Brief Title: Omega-3 Fatty Acids in Preventing Breast Cancer in Women at High Risk of Developing Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000430701; CSMC-00006359; CSMC-00000509
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2006-07

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fatty Acids, Omega-3

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acid

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs or supplements to keep cancer from forming, growing, or coming back. The use of omega-3 fatty acids may prevent breast cancer.

PURPOSE: This randomized clinical trial is studying how well omega-3 fatty acids work in preventing breast cancer in women at high risk of developing breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effects of omega-3 fatty acids on mammographic breast density (MBD) in women at high risk of developing breast cancer.

Secondary

* Determine, preliminarily, the effects of this supplement on cell atypia and breast cell proliferation measured in ductal lavage specimens from these patients.
* Determine the effects of this supplement on circulating hormone and growth factor blood levels in these patients.
* Determine the effects of this supplement on the expression of estrogen-related proteins found in ductal lavage specimens from these patients.
* Determine the effects of this supplement on plasma lipid peroxidation levels in these patients.
* Correlate the modifying effect of lipid peroxidation-related genes with MBD in patients treated with this supplement.

OUTLINE: This is a randomized, pilot study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral placebo three times daily for 12 months.
* Arm II: Patients receive oral omega-3 fatty acids three times daily for 12 months.

In both arms, treatment continues in the absence of the development of ductal carcinoma in situ or invasive carcinoma of the breast or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 80 patients (40 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At increased risk of developing breast cancer, as defined by 1 of the following criteria:

  * 5-year Gail risk ≥ 1.7%
  * Calculated 5-year Gail risk ≥ 5 times the average for age group, as defined by 1 of the following:

    * At least 0.1% (for patients age 20-29)
    * At least 1.0% (for patients age 30-39)
    * At least 1.7% (for patients age 40 and over)
  * Known BRCA1 or BRCA2 mutation carrier
  * Family history consistent with hereditary breast cancer, as defined by any of the following:

    * At least 4 relatives diagnosed with breast cancer at any age
    * At least 2 first-degree relatives diagnosed with breast cancer at age 50 or younger
    * Breast and ovarian cancer diagnosed in the same relative
    * At least 2 occurrences of breast cancer and 1 occurrence of ovarian cancer at any age in the same family
  * Atypical hyperplasia or lobular carcinoma in situ of the breast by prior biopsy
  * History of unilateral ductal carcinoma in situ of the breast
  * History of invasive stage I breast cancer in remission (completed local and systemic standard therapy)
  * History of ovarian cancer in remission for > 5 years
* Baseline mammogram performed within the past 6 months with an interpretation of not suspicious for malignancy (BIRAD 1-3)
* Not eligible for OR refused standard breast cancer risk reduction strategies (e.g., prophylactic oophorectomy, prophylactic mastectomy, or tamoxifen)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* SWOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL

Hepatic

* SGOT and/or SGPT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 2.0 times ULN

Renal

* Creatinine ≤ 2.0 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* No underlying medical, psychiatric, or social condition that would preclude study participation
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* More than 6 months since prior and no concurrent hormonal therapy, including any of the following:

  * Antiestrogens
  * Estrogen
  * Selective estrogen-receptor modulators
  * Progestins
  * Aromatase inhibitors
  * Hormonal contraceptives

Radiotherapy

* Not specified

Surgery

* No prior bilateral mastectomy

Other

* More than 3 months since prior and no concurrent chronic (i.e., > 3 times per week) non-steroidal anti-inflammatory drugs (e.g., aspirin, ibuprofen, or indomethacin) or cyclooxygenase-2 inhibitors
* No prior cancer treatment that would preclude study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-04

PRIMARY OUTCOMES:
Breast density as measured by the Madena method at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, MD, Study Chair — Cedars-Sinai Medical Center
Locations (1):
- Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California, United States